CLINICAL TRIAL: NCT04662125
Title: Comparative Study Between Analgesic Effect of Oral Prednisolone and Oral Pregabalin in Management of Post-dural Puncture Headache in Patients Undergoing Lower Limb Surgeries
Brief Title: Management of Post Dural Pucture Headache After Lower Limb Surgeries: Oral Prednisolone vs Oral Pregabalin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Dina Abdelhameed Elsadek Salem, principal investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6324
Record Dates: First submitted 2020-11-28; First posted 2020-12-10 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Analgesia
Keywords: oral prednisolone; oral pregabalin; post dural puncture headache (PDPH); lower limb surgeries
MeSH Terms: conditions — Agnosia; Post-Dural Puncture Headache | interventions — Caffeine; Acetaminophen; Prednisolone; Pregabalin

STUDY DESIGN:
Intervention Model Description: Analgesic management of post dural puncture headache: oral prednisolone vs oral pregabalin
Who Masked: Participant, Outcomes Assessor
Masking Description: anesthetist not sharing in the study will assess patient
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A (Active Comparator): Group A (conservative treatment): oral fluid intake, recumbent positioning, combination of paracetamol and caffeine tablet three times per day for three days (2 tablets of Panadol-Extra tablet, film coated, GlaxoSmithKline Consumer Healthcare Holdings (US) LLC were given every 8hours) and stool softener and to maintain blinding a tablet of vitamins was given twice per day for three days.
  Interventions: Drug: caffeine, paracetamol tablet
- group B (Active Comparator): Group B (oral prednisolone): patients who received conservative treatment as control group together with oral tablet prednisolone 20 mg once daily plus one tablet of vitamins to maintain blinding for three days.
  Interventions: Drug: Oral prednisolone
- group C (Active Comparator): Group C (oral pregabalin): patients who received conservative treatment as control group together with oral tablet pregabalin 150 mg twice per day for three days.
  Interventions: Drug: oral pregabalin

INTERVENTIONS:
Drug: caffeine, paracetamol tablet — oral fluid intake, recumbent positioning, combination of paracetamol and caffeine tablet three times per day for three days (2 tablets of Panadol-Extra tablet, film coated, GlaxoSmithKline Consumer Healthcare Holdings (US) LLC were given every 8hours) and stool softener and to maintain blinding a tablet of vitamins was given twice per day for three days.
  Arms: group A
Drug: Oral prednisolone — patients who received conservative treatment as control group together with oral tablet prednisolone 20 mg once daily plus one tablet of vitamins to maintain blinding for three days. .
  Arms: group B
Drug: oral pregabalin — patients who received conservative treatment as control group together with oral tablet pregabalin 150 mg twice per day for three days.
  Arms: group C

SUMMARY:
The aim of this study is to compare between oral prednisolone and oral pregabalin in management of PDPH to detect effectiveness of the treatment in reducing severity of PDPH, total rescue analgesic consumption and adverse effects of prednisolone and pregabalin in patients undergoing lower limb surgery.

DETAILED DESCRIPTION:
1. To compare between oral prednisolone and oral pregabalin in reducing severity post-dural puncture headache after spinal anesthesia in patients undergoing lower limb surgeries.
2. To calculate total amount of postoperative analgesic requirement for 72 hours after the onset of the headache in all patient groups.
3. To detect any side effects of the study medications in all patient groups.

ELIGIBILITY:
Inclusion Criteria:

* - Both gender.
* Age: 18- 65 years old.
* Body Mass Index 20-30 kg/m2
* American Society of Anesthesiologist (ASA) physical status I - II.
* Patients are diagnosed as PDPH according to criteria of International Headache Society (IHS) after lower limb surgeries .

Exclusion Criteria:

* - Allergy to study drugs.
* History of chronic headache and migraine.
* History of cerebrovascular accidents and neurological disorders.
* Systemic infection
* History of uncontrolled DM or hepatic disease or pregnant female
* Patient refusal or uncooperative patient.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
pain intensity of headache | From onset of the headache (0 hour).
  measured by Visual Analogue Scale (VAS) on 0-10 cm scale (0-1 no headache, 2-4 mild headache, 5-7 moderate headache and 8-10 sever headache)
pain intensity of headache | at 12 hours
  measured by Visual Analogue Scale (VAS) on 0-10 cm scale (0-1 no headache, 2-4 mild headache, 5-7 moderate headache and 8-10 sever headache)
pain intensity of headache | at 24 hours
  measured by Visual Analogue Scale (VAS) on 0-10 cm scale (0-1 no headache, 2-4 mild headache, 5-7 moderate headache and 8-10 sever headache)
pain intensity of headache | at 48 hours
  measured by Visual Analogue Scale (VAS) on 0-10 cm scale (0-1 no headache, 2-4 mild headache, 5-7 moderate headache and 8-10 sever headache)
pain intensity of headache | at 72 hours
  measured by Visual Analogue Scale (VAS) on 0-10 cm scale (0-1 no headache, 2-4 mild headache, 5-7 moderate headache and 8-10 sever headache)
Headache intensity | From onset of the headache (0 hour).
  modified Lybecker score :1: include patients with mild headache not affecting daily activity with no accompanying symptoms, and oral analgesics work effectively to relieve pain, grade 2: moderate headache that restricts daily activity and leaves the patient in bed for most of the day, injectable analgesia is required to relieve pain, and grade 3: Severe headache with associated symptoms, completely restrict daily activity, with patients kept bed bound for the whole day.
Headache intensity | at 12 hours
  modified Lybecker score :1: include patients with mild headache not affecting daily activity with no accompanying symptoms, and oral analgesics work effectively to relieve pain, grade 2: moderate headache that restricts daily activity and leaves the patient in bed for most of the day, injectable analgesia is required to relieve pain, and grade 3: Severe headache with associated symptoms, completely restrict daily activity, with patients kept bed bound for the whole day.
Headache intensity | at 24 hours
  modified Lybecker score :1: include patients with mild headache not affecting daily activity with no accompanying symptoms, and oral analgesics work effectively to relieve pain, grade 2: moderate headache that restricts daily activity and leaves the patient in bed for most of the day, injectable analgesia is required to relieve pain, and grade 3: Severe headache with associated symptoms, completely restrict daily activity, with patients kept bed bound for the whole day.
Headache intensity | at 48 hours
  modified Lybecker score :1: include patients with mild headache not affecting daily activity with no accompanying symptoms, and oral analgesics work effectively to relieve pain, grade 2: moderate headache that restricts daily activity and leaves the patient in bed for most of the day, injectable analgesia is required to relieve pain, and grade 3: Severe headache with associated symptoms, completely restrict daily activity, with patients kept bed bound for the whole day.
Headache intensity | at 72 hours
  modified Lybecker score :1: include patients with mild headache not affecting daily activity with no accompanying symptoms, and oral analgesics work effectively to relieve pain, grade 2: moderate headache that restricts daily activity and leaves the patient in bed for most of the day, injectable analgesia is required to relieve pain, and grade 3: Severe headache with associated symptoms, completely restrict daily activity, with patients kept bed bound for the whole day.

SECONDARY OUTCOMES:
Associated symptoms of post dural puncture headache | for 72 hours
  The number of participant who has symptoms of post dural pucture headache as nausea, vomiting, diplopia, dizziness and neck stiffness
Adverse effects of the study drugs e.g. sedation, blurred vision, sleepiness, and dizziness | for 72 hours
  In case of sedation, the level will be assessed by using Ramsay Sedation Score (1= anxious or agitated, 2= cooperative and oriented, 3= responds to commands only and 4= brisk response to light tap or loud auditory stimulus)
total dose of rescue analgesia | for 72 hours
  total amount of ketorolac

CONTACTS AND LOCATIONS:
Overall Officials: Dina Salem, MD, Principal Investigator — faculty of medicine , Zagazig university
Locations (1):
- faculty of medicine, Zagazig university, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No